CLINICAL TRIAL: NCT06548282
Title: Efficacy of Acceptance and Commitment Therapy for the Management of Quality of Life in Patients Post Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Sehrish Khan, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2024/88
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Psychological Distress; Type D Personality; Medication Adherence; Quality of Life
MeSH Terms: conditions — Medication Adherence | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Who receives intervention i.e. Acceptance and Commitment Therapy
  Interventions: Other: Acceptance and commitment therapy
- Waitlist Control (Active Comparator): Who would receive intervention after study completion
  Interventions: Other: Acceptance and commitment therapy

INTERVENTIONS:
Other: Acceptance and commitment therapy — Introduction: Build rapport and complete pre-assessment questionnaires.
  First Session:
  Introduce therapist, ACT principles, and MI complications. Provide psychoeducation and assign homework.
  Second Session:
  Review feedback and encourage change. Assign homework.
  Third Session:
  Discuss acceptance and coping strategies. Assign homework.
  Fourth Session:
  Discuss cognitive diffusion and unhelpful thoughts. Assign homework.
  Fifth Session:
  Explore self-concept and mindfulness. Assign homework.
  Sixth Session:
  Identify and elaborate on values. Assign homework.
  Seventh Session:
  Discuss values, goals, and barriers. Assign homework.
  Eighth Session:
  Discuss commitment to action and relapse prevention. Administer post-test and express gratitude.

SUMMARY:
The present study aims to investigate the efficacy of acceptance and commitment therapy for the management of quality of life in patients post-myocardial infarction

DETAILED DESCRIPTION:
The current quantitative study is carried out in two steps. A cross-sectional survey assesses quality of life and associated factors during the first step. A randomized controlled trial will be done during the second step where patients with myocardial infarction who are identified with type D personality characteristics, psychological distress, low level of medication adherence, low social support, low quality of life, low acceptance and psychological flexibility will be randomly assigned to two groups i.e. waitlist control group and intervention group. The acceptance and commitment therapy would be implemented on participants in the interventional group. As the control group is the waitlist control group; initially no intervention will be given to participants in the control group but the intervention will be given to the control group participants once the study is completed.

ELIGIBILITY:
Inclusion Criteria:

1. First-time diagnosed, non-hospitalized patients with myocardial infarction (MI).
2. Patients attending follow-up visits at the hospital.
3. Patients experiencing distress.
4. Patients exhibiting features of Type D personality.
5. Patients reporting low levels of:

   * Quality of Life (QoL)
   * Medication adherence
   * Social support
   * Acceptance
   * Psychological flexibility
6. Patients aged 18 years and above.
7. Both genders.
8. Patients who can understand Urdu.
9. Patients who can provide informed consent.

Exclusion Criteria:

1. Hospitalized patients with myocardial infarction (MI).
2. Patients with myocardial infarction (MI) and other chronic co-morbid diseases, such as:

   * Cancer
   * Cognitive deficits
   * Chronic psychological disorders
3. Patients with silent myocardial infarction.
4. Patients younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Scale Urdu Version | 3 months
  It has 26 items and four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains quality of life and general health items. The minimum value is 26 and the maximum value is 130. Higher scores on the scale indicate higher quality of life and low scores indicate low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sehrish Khan, PhD Scholar, Principal Investigator — Fatima Jinnah women University, Rawalpindi, Pakistan
Locations (2):
- Pakistan (2):
  - Armed Forces Institute of Cardiology, Rawalpindi, Punjab Province
  - Rawalpindi Institute of Cardiology, Rawalpindi, Punjab Province